CLINICAL TRIAL: NCT07038161
Title: Duct To Mucosa Pancreaticojejunostomy (The Novel Modified Cattell Warren Technique) Significantly Reduces POPF: A Single-Center Experience
Brief Title: The Novel Modified Cattell-Warren Duct-To-Mucosa Pancreaticojejunostomy Technique Significantly Reduces POPF.
Acronym: POPF
Status: Completed | Type: Observational
Sponsor: Nepal Medical College and Teaching Hospital (Other)
Responsible Party: Principal Investigator, Nabin Pokharel, Official Title: Prof Dr. Nabin Pokharel, Head of Department of Surgical Gastroenterology Affiliation: Nepal Medical College and Teaching Hospital, Nepal Medical College and Teaching Hospital
Other Study IDs: 45-081/082
Record Dates: First submitted 2025-06-09; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pancreaticoduodenectomy; Distal Pancreatectomy; Postoperative Pancreatic Fistula
Keywords: Duct-to-mucosa; pancreaticojejunostomy; Postoperative pancreatic fistula; Modified Cattell-Warren technique

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Modified Cattell-Warren Technique for Pancreaticojejunostomy: All patients undergoing the duct-to-mucosa (the Modified Cattell-Warren technique) for pancreaticojejunostomy in the Pancreaticoduodenectomy and Distal Pancreatectomy.
  Interventions: Procedure: Modified Cattell-Warren duct-to-mucosa pancreaticojejunostomy; Behavioral: Institutional Prehabilitation Protocol

INTERVENTIONS:
Procedure: Modified Cattell-Warren duct-to-mucosa pancreaticojejunostomy — Technical modification of the original Cattell-Warren technique in all the stitches of both posterior and anterior duct-to-mucosa layer, taking the pancreatic duct with more than 5mm of pancreatic parenchyma adjacent to the duct and towards the jejunal side, taking more than 5 mm of full-thickness jejunum including mucosa.
Behavioral: Institutional Prehabilitation Protocol — Routine perioperative incentive spirometry, four extremities exercise, and nutritional optimization with albumin and Total Parenteral Nutrition

SUMMARY:
Pancreatic surgeries, such as pancreaticoduodenectomy and distal pancreatectomy, are associated with high morbidity and mortality. The most common cause of this morbidity is postoperative pancreatic fistula(POPF). The risk of POPF depends on the texture of pancreatic parenchyma, the size of the main pancreatic duct, and the technique of pancreatic-enteric reconstruction. There are several techniques for pancreaticojejunostomy anastomosis. Among which duct to mucosa is considered a relatively safe anastomosis technique. However, there are several modifications to the duct-to-mucosa technique. The investigators of this study believe that the modified Cattell-Warren duct-to-mucosa technique, which includes taking more than 5 mm of periductal pancreatic parenchyma with the duct and the full-thickness jejunum while performing pancreaticojejunostomy reconstruction with proper perioperative nutritional optimization and prehabilitation, improves patient outcomes. So the investigators aim to assess the risk of POPF in the novel modified Cattell-Warren technique.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is one of the most aggressive malignancies. The incidence of pancreatic cancer is rising, with over 500,000 new cases worldwide, especially with increasing trends in developing countries. It is associated with high morbidity and mortality due to its aggressive nature and late diagnosis of the disease. Only 15-20% of the disease is resectable at presentation, and another 30% of patients have a borderline resectable disease. Pancreaticoduodenectomy (PD) is the only treatment with curative intent for pancreatic head tumors and periampullary tumors. Though the mortality associated with PD has decreased with the experience of surgeons, the morbidity still hovers around 30-50%. Adjuvant chemotherapy is crucial in improving survival outcomes, with median survival reaching 24-30 months. However, a significant subset of patients undergoing PD is unable to undergo or tolerate adjuvant chemotherapy due to its high surgical morbidity, prolonged recovery, or poor performance status. Around 30-40% of patients do not receive adjuvant therapy as planned due to surgical morbidity, which negatively impacts long-term survival.

Pancreatic surgery, including PD and distal pancreatectomy (DP) is a highly complex surgery requiring multiple reconstructive anastomoses with significant risk of postoperative morbidity, even in a high-volume center. Pancreaticojejunostomy (PJ) is the most technically demanding reconstructive anastomosis due to its high risk of anastomotic leaks, resulting in postoperative morbidity. The most common cause of this morbidity is due to Postoperative pancreatic fistula (POPF), while other causes include Post-pancreatectomy hemorrhage (PPH), delayed gastric emptying (DGE), biliary and enteric leaks, pancreatic endocrine and exocrine insufficiency, and wound-related complications. POPF is the most feared and dreadful complication following pancreatic surgery for both benign and malignant pathology. The pancreatic parenchymal texture, duct diameter, and technique of anastomosis of the pancreatic-enteric reconstruction are important factors that influence the formation of POPF. Duct-to-mucosa and its modification, Invagination (Dunking), Binding, or Pancreaticogastrostomy (PG) are techniques for the reconstruction of the pancreatic remnant. The Catell-Warren technique, described in 1956, is the duct to mucosa PJ technique, which is a widely used technique that ensures a secure anastomosis of the pancreatic duct with jejunal mucosa. It is considered to be one of the most precise PJ techniques, which is found to reduce POPF significantly. The secure 2-layer anastomosis, minimization of parenchymal trauma, proper ductal drainage, better healing, and lower risk of anastomotic strictures make this technique an optimal PJ technique. The duct to mucosa PJ technique is the preferred technique when the MPD diameter is > 3mm. However, this technique is being safely done even with an MPD diameter of >1mm without a significant increase in POPF risk. Among various PJ techniques, the duct-to-mucosa technique is widely used because of its precise and direct alignment between the pancreatic remnant and jejunal mucosa, theoretically minimizing the risk of POPF.

However, modification in surgical technique, variation in use of internal or external stents, use of perioperative octreotide, patient-specific factors, and institutional surgical protocol create inconsistent results in clinical practice. Despite the advantages of the duct-to-mucosa PJ technique, the clinical efficacy and safety of this technique remain debated, with some studies suggesting no clear superiority over other methods. Given the ongoing debate and variability in outcomes, there is a need for focused evaluation of the duct-to-mucosa PJ to quantify its impact on the incidence and severity of POPF, technical feasibility, and safety of the technique, and to standardize the anastomotic technique in pancreatic surgery.

Demographic data, investigation parameters, intraoperative findings, and surgical outcomes will be retrieved from the departmental database. Statistical tests for comparison will be done using SPSS version 16.0. Continuous variables will be presented as Mean + Standard Deviation (SD), and categorical variables will be presented as Number (percentage). Analysis will be done using the chi-square test and student t-test wherever applicable, and other statistical tests as per requirement. The level of significance will be set at 5%, and p p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing duct to mucosa PJ (the modified Cattell Warren technique) in pancreatic surgery for presumed or diagnosed malignancy of the head of the pancreas and periampullary carcinoma.
* Patient undergoing distal pancreatectomy for presumed or diagnosed malignancy or cystic neoplasm of the pancreas involving the body and tail.
* Age > 18 years

Exclusion Criteria:

* Other techniques of reconstruction like Dunking, Blumgart's, and binding technique.
* Patient with previous pancreatic resection for any etiology
* Patient undergoing extended pancreaticoduodenectomy
* Arterial resection or divestment
* Multi-visceral resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing the modified Cattell-Warren duct-to-mucosa pancreaticojejunostomy technique in the pancreaticoduodenectomy or distal pancreatectomy in the department of Surgical Gastroenterology in the Nepal Medical College and Teaching Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant postoperative pancreatic fistula | Assessed between postoperative day 3 and up to 30 days
  To assess the rate of clinically relevant postoperative pancreatic fistula (CR POPF) in the standard time frame as per ISGPS guidelines.

SECONDARY OUTCOMES:
Number of patients with other postoperative complications based on the Clavien-Dindo Classification grading | up to 90 postoperative days and during follow-up in OPD (as per departmental protocol for this study)
  Number of patients with other postoperative complications based on the Clavien-Dindo Classification grading in the standard time frame as per ISGPS guidelines
Length of hospital stay | Length of hospital stay (LOS) was defined as the time (in days) from the date of surgery to the date of hospital discharge, assessed up to 90 days postoperatively.
  The association between complication severity and LOS was evaluated by comparing LOS across Clavien-Dindo grades. Prolonged LOS was defined as hospitalization >75th percentile of the cohort.
Mortality | up to 30 postoperative days or till the date of in-hospital mortality due to any cause, assessed upto 30 postoperative days
  Number of patients with in-hospital postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Nabin Pokharel, MBBBS,MS,MCh, Principal Investigator — Nepal Medical College and Teaching Hospital
Locations (1):
- Gonish Hada, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Yu XF, Yao H, Xu S, Ma YQ, Chai C. Safety and feasibility of modified duct-to-mucosa pancreaticojejunostomy during pancreatoduodenectomy: A retrospective cohort study. World J Gastrointest Surg. 2023 Sep 27;15(9):1901-1909. doi: 10.4240/wjgs.v15.i9.1901. PMID 37901736
- [Background] Sun X, Zhang Q, Zhang J, Lou Y, Fu Q, Zhang X, Liang T, Bai X. Meta-analysis of invagination and duct-to-mucosa pancreaticojejunostomy after pancreaticoduodenectomy: An update. Int J Surg. 2016 Dec;36(Pt A):240-247. doi: 10.1016/j.ijsu.2016.11.008. Epub 2016 Nov 5. PMID 27826046
- [Background] Hai H, Li Z, Zhang Z, Cheng Y, Liu Z, Gong J, Deng Y. Duct-to-mucosa versus other types of pancreaticojejunostomy for the prevention of postoperative pancreatic fistula following pancreaticoduodenectomy. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD013462. doi: 10.1002/14651858.CD013462.pub2. PMID 35289922
- [Background] Hao X, Li Y, Liu L, Bai J, Liu J, Jiang C, Zheng L. Is duct-to-mucosa pancreaticojejunostomy necessary after pancreaticoduodenectomy: A meta-analysis of randomized controlled trials. Heliyon. 2024 Jun 15;10(13):e33156. doi: 10.1016/j.heliyon.2024.e33156. eCollection 2024 Jul 15. PMID 39040391